CLINICAL TRIAL: NCT03660917
Title: Riluzole in Patients With Spinocerebellar Ataxia Type 7: a Randomized , Double-blind, Placebo-controlled Pilot Trial With a Lead in Phase
Brief Title: Riluzole in Patients With Spinocerebellar Ataxia Type 7
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Ristori, Principal Investigator, S. Andrea Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIFA-2016-02365063
Record Dates: First submitted 2018-05-15; First posted 2018-09-07 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: SCA7
MeSH Terms: interventions — Riluzole

STUDY DESIGN:
Intervention Model Description: We opted for a randomized, double-blind, placebo-controlled pilot trial with a lead-in phase. Moreover, the patients to be included in the placebo arm will receive riluzole during the last 6 months of study, so that all patients will undergo the active drug in the last phase of the study.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riluzole (Experimental): Riluzole 50 mg twice daily for 12 months in the treated group. In pre-pubertal subjects the dosage will be adjusted on a mg/m2 basis according to the recommended human daily dose (RHDD; 100 mg).
  Interventions: Drug: Riluzole
- Placebo + riluzole (Placebo Comparator): Placebo twice daily for 6 months and riluzole 50 mg twice daily for the following 6 months in the comparison group
  Interventions: Drug: Riluzole; Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — Study drug will be orally dispensed in doses of 50 mg twice daily for 12 months in the treated group.
Drug: Placebo — Placebo drug for 6 months, however they will receive riluzole during the last 6 months of study, so that all patients will undergo the active drug in the last phase of the study.
  Arms: Placebo + riluzole

SUMMARY:
Spinocerebellar ataxia type 7 (SCA7) belongs to the dominant forms of inherited cerebellar ataxias (CA), being one of the rarest form. SCA7 has no therapeutic options, so that the relentless course, the important visual deficit that accompanies CA, and the possibility of disease development in childhood are pressing unmet needs. The investigators published encouraging data on riluzole in inherited CA other than SCA7. These results prompted off-label use of riluzole in single cases of SCA7 in Italy and United States, suggesting possible efficacy of the drug in this condition.

DETAILED DESCRIPTION:
The investigators propose a clinical trial in SCA7 patients performing a serial evaluation of riluzole effects on stringent outcome measures: ophthalmological metrics, scale for the assessment and rating of ataxia (SARA) scores, and safety biomarkers.

The study design will be a randomized , double-blind, placebo-controlled pilot trial with a lead-in phase. The design will include a run-in phase of 6 months for all the participants, assessing ophthalmological metrics and SARA scores at the month 0, 3, and 6. Then one arm will undergo riluzole for other 12 months, while the other will take placebo for 6 months, and riluzole for the following 6 months; from both groups the same evaluations will be obtained at the month 12, 15 and 18 of the study.

Thirty-four patients will be enrolled at 4 clinical Centers (3 in Italy and one in U.S.). The clinical epidemiology aspects (design of the study, statistical analysis and enrollment process) will be followed by National Rare Diseases Centre and Complex Diseases Group of National Centre of Epidemiology, Surveillance and Health Promotion of National Institute of Health.

Eligible subjects for this study are patients (at least 7-year old) with positive genetic test for SCA7. Serious systemic illnesses or conditions (cardiac, haematologic and hepatic diseases) known for enhancing the side effects of riluzole, pregnancy or breastfeeding will be exclusion criteria.

Participants will be randomly assigned (1:1) to riluzole (50 mg twice daily) or placebo. In pre-pubertal subjects the dosage will be adjusted on a mg/m2 basis according to the recommended human daily dose (100 mg).

At baseline and after 3, 6, 12, 15 and 18 months, symptoms, physical and neurological signs, and SARA score will be recorded. At the same time points the following quantitative ophthalmologic assessments will be performed:

* corrected visual acuity (right eye and left eye measurements) expressed as logMAR units with the ETDRS chart (either back-illuminated or projected).
* Color vision via a Farnsworth D15 Arrangement Test.
* Visual evoked potential are elicited using transient Pattern Reversal stimuli and monocular stimulation.
* Electroretinography
* Optical Coherence tomography with macular map of both eyes.
* Computerized visual field examination by standard automated perimetry and kinetic perimetry Every three months electrocardiogram and a laboratory profile will be obtained for drug safety.

The co-primary endpoints will be the proportion of patients with stability of SARA score and visual acuity (in log MAR units) at 18 months, compared to the mean values of t0-t3-t6 evaluations.

A sample size of 17 patients per group (a total of 34 patients) had 80% power and an α value of 10% to detect a difference between the two groups of 35% in the co-primary end points. This calculation took into account published data on riluzole in CA.

Data will be expressed as mean (SD) for continuous variables and as proportions for categorical variables. Comparisons between riluzole and placebo group will be assessed using the t test for unpaired data for continuous variables and odds ratio with a relative 95% CI for categorical data. An intention-to-treat analysis will be done adopting a last observation carried forward method. A logistic regression model will be done at 18 months to adjust the results for the main baseline characteristics; p values less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* positive genetic test for SCA7.

Exclusion Criteria:

* cardiac arrhythmias;
* haematologic diseases;
* hepatic diseases with serum values of alanine aminotransferase, aspartate aminotransferase or bilirubin > 1·5 times above normal limit;
* pregnancy (women of childbearing potential agreed to use contraception);
* breastfeeding.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
visual acuity expressed as log MAR units | 18 months
  the metric to quantify the best corrected visual acuity, by applying the ETDRS chart (either back-illuminated or projected) with the patient's correction for distance
the proportion of patients with stable Scale for the assessment and rating of ataxia (SARA) score | 18 months
  neurological assessment for ataxia. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia). When completing the outcome measure each category is assessed and scored accordingly. Scores for the eight items range as follows:
  Gait (0-8 points), Stance (0-6 points), Sitting (0-4 points) Speech disturbance (0-6 points) Finger chase (0-4 points) Nose-finger test (0-4 points) Fast alternating hand movement (0-4 points) Heel-shin slide (0-4 points) Once each of the 8 categories have been assessed, the total is calculated to determine the severity of ataxia.
  For motor activities of the four extremities (items 5-8), assessments are performed bilaterally, and the mean values are used to obtain the total score.

SECONDARY OUTCOMES:
Farnsworth D15 Arrangement Test | 18 months
  quantitative ophthalmologic assessments
Visual evoked potentials | 18 months
  quantitative ophthalmologic assessments
Electroretinography | 18 months
  quantitative ophthalmologic assessments
Optical Coherence tomography | 18 months
  quantitative ophthalmologic assessments
Scale for the assessment and rating of ataxia (SARA) score | 18 months
  neurological assessment for ataxia. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia). When completing the outcome measure each category is assessed and scored accordingly. Scores for the eight items range as follows:
  Gait (0-8 points), Stance (0-6 points), Sitting (0-4 points) Speech disturbance (0-6 points) Finger chase (0-4 points) Nose-finger test (0-4 points) Fast alternating hand movement (0-4 points) Heel-shin slide (0-4 points) Once each of the 8 categories have been assessed, the total is calculated to determine the severity of ataxia.
  For motor activities of the four extremities (items 5-8), assessments are performed bilaterally, and the mean values are used to obtain the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurological Unit, S. Andrea Hospital, Faculty of Medicine and Psychology, "Sapienza" University of Rome, Rome, Italy